CLINICAL TRIAL: NCT02952157
Title: Effect on Postoperative Sore Throat of Lidocaine Jelly Application Over the Endotracheal Tube of Tapered-shaped Cuff
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LidoTaper
Record Dates: First submitted 2016-10-20; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Sore Throat
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Sham Comparator): Normal saline will be applied to the endotracheal tube.
  Interventions: Drug: Normal saline application
- Lidocaine (Active Comparator): Lidocaine jelly will be applied to the endotracheal tube.
  Interventions: Drug: Lidocaine jelly application

INTERVENTIONS:
Drug: Lidocaine jelly application
  Arms: Lidocaine
Drug: Normal saline application
  Arms: Control

SUMMARY:
Postoperative sore throat is a complication after general anesthesia requiring endotracheal intubation. The investigators will evaluate the efficacy of lidocaine jelly application on the endotracheal tube with taper-shaped cuff regarding postoperative sore throat.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Patients scheduled for general anesthesia with endotracheal intubation
* Patients scheduled for surgery which duration is expected to less than 3 hr

Exclusion Criteria:

* Difficult airway
* Rapid sequence induction
* Recent sore throat
* Recent upper respiratory infection
* Asthma
* Chronic obstructive pulmonary disease
* Chronic cough
* Pregnancy
* Allergy to lidocaine
* Friable teeth
* History of head and neck surgery
* Multiple intubation attempts
* Regional anesthetic agents
* Gastric tube
* Dexamethasone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2016-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with sore throat | At 24 hr

SECONDARY OUTCOMES:
Number of participants with sore throat | At 1, 6, and 12 hr
Number of participants with hoarseness | At 1, 6, 12 and 24 hr
Number of participants with throat numbness | At 1, 6, 12 and 24 hr
Number of participants with nausea | At 1, 6, 12 and 24 hr
Number of participants with vomiting | At 1, 6, 12 and 24 hr
Number of participants with cough | At 1, 6, 12 and 24 hr
Number of participants with dry mouth | At 1, 6, 12 and 24 hr
Number of participants with additional pain medication | At 24 hr

IPD SHARING:
Plan to Share IPD: No